CLINICAL TRIAL: NCT02012517
Title: Antibiotic Prophylaxis in Prosthetic Breast Reconstructions
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Yasmin Maor, Head of the infectious didease service to the hospitalized patient, infectious disease unit, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0447-13-SMC
Record Dates: First submitted 2013-12-05; First posted 2013-12-16 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Surgical Site Infections
Keywords: surgical site infection; breast reconstruction; drains; prophylaxis
MeSH Terms: conditions — Surgical Wound Infection | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- short antibiotic course (Active Comparator): Intravenous 2 gram cefazolin every 8 hours for 24 hours beginning at surgery
  Interventions: Drug: Short antibiotic course (standard of care)
- Prolonged antobiotic treatment (Experimental): Intravenous 2 gram cefazolin every 8 hours for 48 hours starting at surgery followed by oral cefalexin 500 mg every 6 hours until removal of drains
  Interventions: Drug: Prolonged antibiotic treatment

INTERVENTIONS:
Drug: Prolonged antibiotic treatment
  Other Names: Intravenous cefazolin 2 grams every 8 hours for 48 hours starting at surgery followed by oral cefalexin 500 mg every 6 hours until removal of drains
  Arms: Prolonged antobiotic treatment
Drug: Short antibiotic course (standard of care)
  Other Names: Intravenous cefazolin 2 grams every 8 hours for 24 hours starting at surgery
  Arms: short antibiotic course

SUMMARY:
The added benefit of prolonged antibiotic prophylactic treatment in patients undergoing breast reconstruction who have drains placed for several days after surgery is controversial. In this study we aim to compare two prophylactic regimens: 1. 24 hour antibiotic treatment prior to surgery with cefazolin 2. a prolonged antibiotic regimen consisting of 48 hours cefazolin treatment followed by oral therapy with cephalexin until the removal of the drains. Patients will sign an informed consent form prior to the surgery and will be randomized to one of the antibiotic regimens. Patients will be closely followed up to one year after surgery. The number of surgical site infections according to the NNIS criteria and loss of breast implants will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

All criteria should be present:

1. Signing an informed consent form
2. Reconstructive breast surgery
3. One drain or more remained after surgery -

Exclusion Criteria:

Age < 18 years Active infection at the surgical site at the operation time or in close proximity to the surgical site Immune deficiency state

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
surgical site infection | 1 year
  The percentage and number of surgical site infections assessed according to the NNIS criteria up to one year after reconstructive breast surgery will be compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Maor, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Department of plastic surgery, Sheba medical center, Tel Litwinsky, Israel